CLINICAL TRIAL: NCT07311317
Title: Assessment of the Accuracy of a Novel Cellular-Level Fluorescence-Guided Imaging Technique in Scanning Tumor Margins During Breast Tumor Resection: A Prospective, Self-Controlled Study
Brief Title: Cellular-Level Fluorescence Imaging for Intraoperative Margin Assessment in Breast Cancer
Acronym: FLASH
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: West China Fourth Hospital, Sichuan University (Unknown); The Fourth People's Hospital of Sichuan Province (Unknown)
Responsible Party: Principal Investigator, Du Zhenggui, deputy director of breast center, West China Hospital
Other Study IDs: 2025-1955
Record Dates: First submitted 2025-12-02; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Breast Cancer,; Fluorescence-guided; Cellular
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Accurate intraoperative margin assessment in breast cancer surgery remains challenging. Current reliance on frozen section pathology is limited by prolonged processing time, sampling constraints, and resource intensity, contributing to variable outcomes.

The EndoSCell Scanner is a novel cellular-resolution fluorescence-guided imaging technology designed to address these limitations. It enables real-time, pathology-level visualization of malignant cellular features at the surgical bed. With a 3mm probe allowing comprehensive 360° margin assessment, it reduces procedural time to under five minutes and may significantly lower secondary surgery rates.

This prospective, self-controlled study aims to evaluate the accuracy of the EndoSCell Scanner for intraoperative margin assessment in patients undergoing mastectomy. Its performance will be systematically compared against both frozen section and final paraffin pathology to validate sensitivity and operational efficiency. If proven effective, this technology could become a standard adjunct tool, standardizing precision in breast cancer surgery and improving patient outcomes by enhancing surgical consistency.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, self-controlled study. Basis for Sample Size Calculation: According to the results of the first phase, the accuracy of frozen pathology is 98.2%. Assuming that the detection interpretation results of ES are not inferior to intraoperative frozen pathology, a one-sided test will be conducted, with α=0.02, 1-β=0.8, and the non-inferiority margin is 0.02. The estimated required sample size is 593. Considering a 10% exclusion rate, the total sample size will be 659. Each patient is expected to have at least 4 samples taken, totaling 165 patients.

Data Collection:1)Basic patient information: age, gender; 2)Tumor diagnosis (including imaging diagnosis): location, size, and staging; 3)Intraoperative collected information: surgery start time, surgery end time; 4)Training and testing records of the physicians in the ES interpretation group; 5)Interpretation records: a.ES start time, ES interpretation end time, ES interpretation results, ES image satisfaction; b.Frozen pathology submission time, report receipt time, report results; c.Paraffin pathology submission time, report time, and report results.

The statistical analysis will be performed using SAS statistical software, version 9.4 or higher. All statistical tests will be two-sided. A P value less than or equal to 0.05 will be considered statistically significant. The description of quantitative indicators will include the mean, standard deviation, median, minimum, maximum, and interquartile range. The description of categorical indicators will use the number and percentage of each category. The comparison of general conditions between the two groups will be analyzed using appropriate methods based on the type of indicators. The consistency evaluation of quantitative data will use the Bland-Altman method and ICC.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 70 years
* Patients scheduled for breast tumor resection
* Clinically or radiologically showing a solitary lesion and

  1. (Before neoadjuvant chemotherapy) Maximum tumor diameter ≤ 5cm;
  2. cN0-1;
  3. No clinical or imaging evidence of nipple, skin, chest wall invasion, or distant metastasis before surgery.
* Subjects voluntarily sign informed consent or are exempted from signing upon approval by the ethics committee.

Exclusion Criteria:

* Inflammatory breast cancer;
* Patients allergic to methylene blue and sodium fluorescein;
* Unable to understand the trial requirements or unable to complete the study follow-up plan;
* Pregnant and breastfeeding women;
* Patients unable to complete follow-up due to mental illness, cognitive or emotional disorders;
* Those with severe comorbidities (such as organ dysfunction, immune deficiency) or poor general condition;
* Those participating in other clinical studies that may affect this trial;
* Those for whom satisfactory specimens for both frozen pathology and paraffin pathology cannot be obtained during surgery;
* Those who cannot obtain a paraffin pathology report.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll 165 adult female patients scheduled to undergo breast surgery for histologically confirmed breast cancer. Eligible participants must provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the sensitivity and specificity of the EndoSCell Scanner (ES) detection, using paraffin pathology as the gold standard, in comparison to rapid frozen section (FS) pathology. | 3 month

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - the Fourth People'S Hospital of Sichuan Province, Chengdu
  - West China Fourth Hospital, Sichuan University, Chengdu
  - West China Hospital, Chengdu

IPD SHARING:
Plan to Share IPD: Undecided